CLINICAL TRIAL: NCT04256928
Title: The Effect of Hair Removal on Intraoperative Contamination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Ditte Harder, Principal Investigator, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 70136
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Intraoperative Complications
MeSH Terms: conditions — Intraoperative Complications

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the intervention group (preoperative electrical clipping) clipping or the control group (leaving the body hair intact) using a 1:1 randomization ratio. The randomization is performed electronically by a medical student or the operating surgeon and the pre-assessment consultation.
  Hair removal is performed with an electric clipper. Clipping is performed by hospital staff on the day of surgery. The degree of body hair on both knees is photo-documented for all participants, for the intervention group after the clipping of body hair on the relevant knee has been performed.
  4 microbiological samples will be taken during surgery from each participant using Copan ESwabs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group of participants will have any body hair in the operative field clipped with an electrical clipper by hospital personnel, during preparation for planned surgery.
  4 microbiological samples will be taken from all participants in this group.
  Interventions: Procedure: Preoperative electrical clipping
- Control group (No Intervention): This group of participants serve as the control group. Any body hair in the operative field is left intact.
  4 microbiological samples will be taken from all participants in this group.

INTERVENTIONS:
Procedure: Preoperative electrical clipping — Body hair in the operative field will be clipped with an electrical clipper by hospital personnel during preparation to planned surgery.
  Arms: Intervention group

SUMMARY:
A prospective, non-blinded, randomized controlled trial with the purpose of investigating, whether preoperative electrical clipping of body hair affects the risk of intraoperative contamination.

The primary investigators hypothesis is this: Preoperative electrical clipping of body hair in the operative field lowers the risk of intraoperative contamination.

200 male participants, 18 years or older, with a planned primary knee replacement surgery, will be enrolled.

During surgery, four microbiological samples will be taken from each participant.

The primary outcome is whether there is intraoperative contamination of the surgical site or not, determined by identification of any grown bacteria from the samples.

If this study finds, that the contamination rate is lowered by preoperative electrical clipping of body hair, it will provide a cost-effective method of reducing the risk of intraoperative contamination and consequent postoperative infection, a solid argument for a change of current guidelines for preoperative hair removal, and provide additional information pointing towards body hair as a possible explanation for the increased infection rate in men.

DETAILED DESCRIPTION:
A late ph.d.-study conducted at Herlev and Gentofte Hospital has shown a 15 percentage difference in contamination rates when comparing participants who had their body hair removed preoperatively, and those who did not.

Based on the finds in the aforementioned study, the hypothesis for this study is that preoperative electrical clipping of body hair in the operative field lowers the risk of intraoperative contamination.

The purpose of this study is to investigate, whether preoperative electrical clipping of body hair affects the risk of intraoperative contamination.

A prospective, non-blinded, randomized controlled trial will be performed. The study population consists of 200 male patients, 18 years or older, with a planned primary knee replacement surgery. The study population consists of only male patients, since males generally have denser body hair and a higher contamination rate than females. Exclusion criteria include known skin disease, use of antibiotics 4 weeks prior to surgery, if patients due to mental reasons, a language barrier or other reasons are unable to participate in the study, as well as no body hair in the surgical field.

Participants will be randomized to either the intervention group (preoperative electrical clipping) or the control group (leaving the body hair intact) using a 1:1 randomization ratio. The randomization is performed electronically by a medical student or the operating surgeon and the pre-assessment consultation.

Clipping is performed by hospital staff on the day of surgery. The degree of body hair on both knees is photo-documented for all participants, for the intervention group after the clipping of body hair on the relevant knee has been performed.

During the surgery, biological material from every participant is collected as four microbiological samples, taken using Copan ESwabs. The first swab is taken before the skin is surgically prepared, the second immediately after incision of the skin, the third swab is taken just prior to the change of gloves performed before cementation of the prothesis, and the last swab is taken after closure of the joint capsule before closure of the skin. Samples will be collected at Orthopedic Departments of Gentofte Hospital. All samples will be sent to Department of Clinical Microbiology, Herlev Hospital, for culturing.The bacteria will be identified following Danish guidelines.

The material consists of culture results from all samples. The primary outcome is whether there is intraoperative contamination of the surgical site or not. This is determined by identification of any grown bacteria.The material will be statistically analyzed using the program R Studio. Since data is categorial, a chi-squared test will be performed to evaluate the significance of the possible difference of contamination rate in the two participant groups.

All possibilities for conducting the study are known to exist, as the method described above has previously been used in the PhD study conducted at the department: "Intraoperative microbial contamination, its prevention and its consequences for outcomes following knee replacement surgery- The ICON study".

Personal data is processed as part of the project. All handling and processing of personal data follows the Data Protection Regulation and the Data Protection Act.

Data collected during the pre-assessment consultation will be entered directly into a database. Only data in this database will be available to the investigators conducting the study, for further analysis. Information about the microbiological samples and cultures will be entered into the database as well. All information in the database will be anonymized 2 years after collection of data is complete.

By consenting to participating in this study, participants also consent to the investigators conducting the study, Herlev-Gentofte Hospital and their representatives to be given direct access to the collected data. Consenting to participate also involves consenting that the Regional Committee on Health Research Ethics are allowed direct access to all data collected, to facilitate their control with the project.

If this study finds, that the contamination rate is lowered by preoperative electrical clipping of body hair, it will not only provide a cost-effective method to reduce the risk of intraoperative contamination and consequent postoperative infection, but may also lead to a change of current guidelines to preoperative electrical clipping of body hair becoming a permanent practice. In addition, the study will confirm existing finds pointing towards body hair as a possible explanation for the increased infection rate in men.

A decrease in the incidence of infections will save patients from unpleasant and often prolonged consequences of infection, including pain, revisions, antibiotic treatments and, at worst, loss of mobility. In addition, fewer infections will lead to savings in the health care system, with the release of funds and beds, to the benefit of patients in general and the social economy.

ELIGIBILITY:
Inclusion Criteria:

* Planned primary knee replacement surgery

Exclusion Criteria:

* Known skin disease
* Use of antibiotics 4 weeks prior to surgery
* If patients due to mental reasons, a language barrier or other reasons are unable to participate in the study
* No body hair in the surgical field

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study population consists of only males, since males generally have denser body hair and a higher contamination rate than females.
Enrollment: 200 (Estimated)
Dates: Start 2020-02-15 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative contamination rate | 1 year
  Rate of contamination as amount of indentified bacteria cultured.

CONTACTS AND LOCATIONS:
Overall Officials: Ditte Harder, Student, Principal Investigator — Herlev og Gentofte Hospital, Ortopædkirurgisk Afdeling T
Locations (1):
- Ortopædkirurgisk Afdeling T, Herlev og Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual partcipant data, but anonymized data can be made available upon request after publication of the study.

REFERENCES:
- [Background] Hesselvig AB, Bjarnsholt T, Arpi M, Madsen F, Odgaard A, group ObotIs. The use of iodine impregnated incision drape in knee arthroplasty surgery - a prospective, randomized trial.
- [Background] Gallo J, Kolar M, Novotny R, Rihakova P, Ticha V. Pathogenesis of prosthesis-related infection. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2003 Nov;147(1):27-35. doi: 10.5507/bp.2003.004. PMID 15034602
- [Background] Byrne AM, Morris S, McCarthy T, Quinlan W, O'byrne JM. Outcome following deep wound contamination in cemented arthroplasty. Int Orthop. 2007 Feb;31(1):27-31. doi: 10.1007/s00264-006-0121-z. Epub 2006 Apr 4. PMID 16586132
- [Background] Jonsson EO, Johannesdottir H, Robertsson O, Mogensen B. Bacterial contamination of the wound during primary total hip and knee replacement. Median 13 years of follow-up of 90 replacements. Acta Orthop. 2014 Apr;85(2):159-64. doi: 10.3109/17453674.2014.899848. PMID 24650025
- [Background] Al-Maiyah M, Hill D, Bajwa A, Slater S, Patil P, Port A, Gregg PJ. Bacterial contaminants and antibiotic prophylaxis in total hip arthroplasty. J Bone Joint Surg Br. 2005 Sep;87(9):1256-8. doi: 10.1302/0301-620X.87B9.15685. PMID 16129753
- [Background] Webster J, Alghamdi A. Use of plastic adhesive drapes during surgery for preventing surgical site infection. Cochrane Database Syst Rev. 2015 Apr 22;2015(4):CD006353. doi: 10.1002/14651858.CD006353.pub4. PMID 25901509
- [Background] Falk-Brynhildsen K, Friberg O, Soderquist B, Nilsson UG. Bacterial colonization of the skin following aseptic preoperative preparation and impact of the use of plastic adhesive drapes. Biol Res Nurs. 2013 Apr;15(2):242-8. doi: 10.1177/1099800411430381. Epub 2012 Jan 24. PMID 22278031
- [Background] Grice EA, Kong HH, Renaud G, Young AC; NISC Comparative Sequencing Program; Bouffard GG, Blakesley RW, Wolfsberg TG, Turner ML, Segre JA. A diversity profile of the human skin microbiota. Genome Res. 2008 Jul;18(7):1043-50. doi: 10.1101/gr.075549.107. Epub 2008 May 23. PMID 18502944
- [Background] Arnold WV, Shirtliff ME, Stoodley P. Bacterial biofilms and periprosthetic infections. Instr Course Lect. 2014;63:385-91. PMID 24720323
- [Background] Aboltins C, Daffy J, Choong P, Stanley P. Current concepts in the management of prosthetic joint infection. Intern Med J. 2014 Sep;44(9):834-40. doi: 10.1111/imj.12510. PMID 24942508
- [Background] Trampuz A, Zimmerli W. Prosthetic joint infections: update in diagnosis and treatment. Swiss Med Wkly. 2005 Apr 30;135(17-18):243-51. doi: 10.4414/smw.2005.10934. PMID 15965826
- [Background] Lange-Asschenfeldt B, Marenbach D, Lang C, Patzelt A, Ulrich M, Maltusch A, Terhorst D, Stockfleth E, Sterry W, Lademann J. Distribution of bacteria in the epidermal layers and hair follicles of the human skin. Skin Pharmacol Physiol. 2011;24(6):305-11. doi: 10.1159/000328728. Epub 2011 Jul 15. PMID 21757977
- [Background] Jose B, Dignon A. Is there a relationship between preoperative shaving (hair removal) and surgical site infection? J Perioper Pract. 2013 Jan-Feb;23(1-2):22-5. doi: 10.1177/1750458913023001-203. PMID 23413532
- [Background] Pan A, Ambrosini L, Patroni A, Soavi L, Signorini L, Carosi G, Santini C; Gruppo Italiano di Studio sulle Infezioni in Cardiochirurgia Study Group. Adherence to surgical site infection guidelines in Italian cardiac surgery units. Infection. 2009 Apr;37(2):148-52. doi: 10.1007/s15010-008-7474-8. Epub 2009 Mar 23. PMID 19308319
- [Background] Broekman ML, van Beijnum J, Peul WC, Regli L. Neurosurgery and shaving: what's the evidence? J Neurosurg. 2011 Oct;115(4):670-8. doi: 10.3171/2011.5.JNS102003. Epub 2011 Jul 1. PMID 21721875
- [Background] Lefebvre A, Saliou P, Lucet JC, Mimoz O, Keita-Perse O, Grandbastien B, Bruyere F, Boisrenoult P, Lepelletier D, Aho-Glele LS; French Study Group for the Preoperative Prevention of Surgical Site Infections. Preoperative hair removal and surgical site infections: network meta-analysis of randomized controlled trials. J Hosp Infect. 2015 Oct;91(2):100-8. doi: 10.1016/j.jhin.2015.06.020. Epub 2015 Aug 4. PMID 26320612
- [Background] Kjonniksen I, Andersen BM, Sondenaa VG, Segadal L. Preoperative hair removal--a systematic literature review. AORN J. 2002 May;75(5):928-38, 940. doi: 10.1016/s0001-2092(06)61457-9. PMID 12063942
- [Background] Shi D, Yao Y, Yu W. Comparison of preoperative hair removal methods for the reduction of surgical site infections: a meta-analysis. J Clin Nurs. 2017 Oct;26(19-20):2907-2914. doi: 10.1111/jocn.13661. Epub 2017 Mar 12. PMID 27875033
- [Background] Tanner J, Woodings D, Moncaster K. Preoperative hair removal to reduce surgical site infection. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD004122. doi: 10.1002/14651858.CD004122.pub3. PMID 16856029
- [Background] Wilson VanVoorhis CR, Morgan BL. Understanding Power and Rules of Thumb for Determining Sample Sizes. Tutorials in Quantitative Methods for Psychology. 2007;3:43-50.